CLINICAL TRIAL: NCT04368234
Title: Duke Shared Data and Specimen Repository Regarding COVID-19 Patients
Brief Title: Duke COVID-19 Shared Data and Specimen Repository
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105316
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Data Specimen Repository
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biological specimens may include, but are not limited to, tissue, blood, urine, sputum, feces, genetic, and/or cell samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patients: Any Duke patient that is being treated for COVID-19.

SUMMARY:
The purpose of this data repository is to provide a secure and centralized storage location and resource for the collection of essential data and medical specimens, across COVID-19 related protocols at Duke.

DETAILED DESCRIPTION:
The aim of this data repository is to provide a secure and centralized storage location and resource for the collection of core variables of interest, as well as the retaining of relevant patient samples, across COVID-19 related protocols at Duke. The core data variables were in-part selected to specifically match those agreed upon by Academic Medical Centers across the U.S., with the intention of aiding the efficiency and effectiveness of de-identified data reuse for population-level research. An additional benefit is that centralized, shared data storage of demographic and longitudinal variables will reduce subject burden, as many questions will now only need to be asked once, rather than each time a given subject joins another COVID-19 related study at Duke.

This shared data and bio-repository project will house all the core data for all patients with COVID-19 (or suspected cases), as well as individual participants ICFs for all other participating COVID-19 studies enrolling Duke patients. Each participating study will have its own separate IRB approved protocol. Samples may be either collected specifically by the protocol, or include left-over clinical samples from the testing and treatment of patients with COVID-19 at Duke.

ELIGIBILITY:
Subjects will be included in this data repository if they meet the enrollment criteria of any linked/participating IRB-approved protocol, or if they are not enrolled in another COVID-related study but meet one of the following inclusion criteria:

1. Suspected novel Coronavirus (nCoV) infection (Person Under Investigation) and/or
2. Laboratory proven acute novel Coronavirus (nCoV) infection and/or
3. Primary admitting diagnosis of nCoV infection

Studies will include:

* Any COVID-19 clinical research studies recruiting Duke patients
* Excludes: protocols sharing non-consented EHR data with national/international repositories and studies that are recruiting community participants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any Duke patient that is receiving treatment for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Development of data repository to provide a secure, centralized storage location for COVID-19 related specimens | Up to 5 years
  This shared data and bio-repository project will house all the core data for all patients with COVID-19 (or suspected cases), as well as individual participant's Informed Consent Forms for all other participating COVID-19 studies enrolling Duke patients. Each participating study will have its own separate IRB approved protocol. Samples may be either collected specifically by the protocol, or include left-over clinical samples from the testing and treatment of patients with COVID-19 at Duke.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Woods, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No